CLINICAL TRIAL: NCT01621880
Title: Effect of Bevacizumab on Radiation-induced Brain Necrosis in Patients With Nasopharyngeal Carcinoma
Acronym: BRAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012025; SYSN001 (Other: Sun Yat-sen Memorial Hospital, Neurology department)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Nasopharyngeal Carcinoma; Adverse Effect of Radiation Therapy; Brain Necrosis
Keywords: radiation-induced brain necrosis; nasopharyngeal carcinoma; Bevacizumab; Methylprednisolone
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Radiation Injuries | interventions — Bevacizumab; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Active Comparator): Patients receive bevacizumab 5mg/kg intravenously over 30-90 minutes on day1. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bevacizumab
- Corticosteroid (Active Comparator): Patients in the corticosteroid group were treated with intravenous pulsed-steroid therapy: methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: bevacizumab — Patients receive bevacizumab 5mg/kg intravenously over 30-90 minutes on day1. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Bevacizumab（Avastin）
  Arms: Bevacizumab
Drug: Corticosteroid — Patients in the corticosteroid group were treated with intravenous pulsed-steroid therapy: methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
  Other Names: methylprednisolone
  Arms: Corticosteroid

SUMMARY:
Bevacizumab may have a better effect on brain necrosis caused by radiotherapy.This randomized trial aims to investigate whether bevacizumab may alleviate radiation-induced brain necrosis in patients with nasopharyngeal carcinoma. The effect will be compared with outcomes in patients receiving steroid therapy.

DETAILED DESCRIPTION:
Radiation-induced brain necrosis is a severe complication of radiotherapy in patients with Nasopharyngeal carcinoma. Current neuroprotective therapies show limited benefit in ameliorating this complication of radiotherapy. This study is a randomized, single blind clinical study. The primary aim of this study is to determine whether bevacizumab can alleviate radiation-induced brain necrosis in patients with nasopharyngeal carcinoma, and to compare the treating effect between bevacizumab and steroid.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received radiotherapy for histologically confirmed nasopharyngeal carcinoma.
* Prior irradiation >/= 6 months prior to study entry.
* Radiographic evidence to support the diagnosis of radiation-induced brain necrosis without tumor recurrence.
* Age>/= 18 years. Because on dosing or adverse event data are currently not available on the use of bevacizumab in patients <18years old.
* No prior bevacizumab therapy.
* No evidence of very high intracranial pressure that suggests brain hernia and needs surgery.
* Fertile women who are willing to take contraception during the trial.
* Routine laboratory studies with bilirubin </=upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) < ULN, creatinine <ULN, red-cell count >/= 4,000 per cubic millimeter; white-cell count >/=1500 per cubic millimeter, platelets >/= 75,000 per cubic millimeter; Hb >/=9.0. PT, APTT, INR in a normal range.
* If with history of seizures, patients should be on anticonvulsant therapy. However, preference will be enzyme-non-inducing anticonvulsants.
* Ability to understand and willingness to sign a written informed consent document.
* The patient has no active bleeding or pathological condition that carries a high risk of bleeding; there is no evidence of serious or non-healing wound, ulcer or bone fracture.

Exclusion Criteria:

* Patients with any of the following should be excluded: 1) evidence of metastatic disease; 2)evidence of tumor invasion to major vessels(e.g. the carotid); 3) history of bleeding related to tumor or radiotherapy during or after the completion of radiation.
* Evidence of active central nervous system hemorrhage.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to study enrollment.
* inadequately controlled hypertension (systolic blood pressure (SBP) > 140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg despite antihypertensive medication)
* Severe complications: 1) History of large vessel cerebrovascular accident (CVA) within 6 months; 2) Myocardial infarction or unstable angina within 6 months; 3) New York heart association grade II or greater congestive heart failure; 4) Serious and inadequately controlled cardiac arrhythmia; 5) Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection); 6) Clinically significant peripheral vascular disease; 7) severe infection.
* Evidence of bleeding diathesis or coagulopathy.
* Patients who have received steroid therapy for radiation-induced brain necrosis before the study.
* History of anaphylactic response to bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Ph.D, Principal Investigator — Department of Neurology, Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Luo S, Lai S, Wu Y, Hong J, Lin D, Lin S, Huang X, Xu X, Weng X. Cost-effectiveness analysis of bevacizumab for cerebral radiation necrosis treatment based on real-world utility value in China. Strahlenther Onkol. 2024 Sep;200(9):805-814. doi: 10.1007/s00066-024-02242-6. Epub 2024 Jun 3. PMID 38829437
- [Derived] Xu Y, Rong X, Hu W, Huang X, Li Y, Zheng D, Cai Z, Zuo Z, Tang Y. Bevacizumab Monotherapy Reduces Radiation-induced Brain Necrosis in Nasopharyngeal Carcinoma Patients: A Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2018 Aug 1;101(5):1087-1095. doi: 10.1016/j.ijrobp.2018.04.068. Epub 2018 May 2. PMID 29885994

RESULTS

PARTICIPANT FLOW:
Groups:
- Corticosteroid: Patients in the corticosteroid group were treated with methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
  Corticosteroid: Patients in the corticosteroid group were treated with intravenous pulsed-steroid therapy: methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
Period: Overall Study
Arm/Group | Bevacizumab | Corticosteroid
Started | 58 | 54
Completed | 48 | 49
Not Completed | 10 | 5
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Corticosteroid: Patients in the corticosteroid group were treated with methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
  Corticosteroid: Patients in the corticosteroid group were treated with methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Corticosteroid | Total
Number analyzed (Participants) | 58 | 54 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (7.0) | 50.5 (8.6) | 50.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  China | 58 | 54 | 112
Conventional radiotherapy [Count of Participants; unit: Participants] | 41 | 36 | 77
IMRT(intensity modulated radiation therapy) [Count of Participants; unit: Participants] | 17 | 18 | 35
Dose of nasopharyngeal radiation [Mean (Standard Deviation); unit: Gy] | 69.4 (5.2) | 71.1 (2.4) | 70.3 (4.1)
Dose of neck radiation [Mean (Standard Deviation); unit: Gy] | 58.9 (8.1) | 40.7 (10.3) | 49.7 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment Response
Description: The primary outcome of the trial was the treatment response rate at two months. The definitions of response and progressive disease were based on both the radiographic changes and clinical symptoms. We defined response as both (1)a reduction in edema volume on FLAIR images by ≥25% and (2)no deteriorating symptoms. Progressive disease was defined as either (1)larger than 10% increase in the volume of the lesions; (2)appearance of any new lesion/site; or (3)clear clinical worsening.
Time Frame: At 2 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Corticosteroid
Number analyzed (Participants) | 58 | 54
Participants | 38 | 17

2. Secondary Outcome: Percentage Change in Radiological Measures of Lesion Volume
Description: T1 post-gadolinium imaging was used to measure the enhancement and T2-weighted FLAIR to measure the edema. For lesion measurements, radiologists used manual and semiautomatic approaches to identify the outline of the lesion, and the total volume was estimated with Volume Viewer 2 software(GE Healthcare, AW Suite2.0 6.5.1.z).
Time Frame: Change from baseline to evaluation at 2 months.
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Corticosteroid: Patients in the corticosteroid group were treated methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
  Corticosteroid: Patients in the corticosteroid group were treated with intravenous pulsed-steroid therapy: methylprednisolone 500 mg daily intravenously for three consecutive days followed by oral prednisone 60 mg for five days and gradually tapered 15mg every 5 days. When the prednisone dose reached 30mg per day, it was tapered down more slowly (tapered 5mg every week), until a maintenance dose of 10mg per day was reached. The entire intervention lasted two months. At 2 months, prednisone was stopped.
Arm/Group | Bevacizumab | Corticosteroid
Number analyzed (Participants) | 48 | 49
percentage
  Percentage Change in FLAIR | -51.8 (39.9) | -19.3 (42.5)
  Percentage Change in enhancement | -25.5 (45.2) | -5.0 (44.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of randomization to 6 months after treatment.
Arm/Group | Bevacizumab | Corticosteroid
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/54
Other Adverse Events (participants affected / at risk) | 25/58 | 26/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=58) | Corticosteroid (N=54)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=58) | Corticosteroid (N=54)
Hypertension (Cardiac disorders) | 12 (12) | 10 (10)
Fatigued (General disorders) | 7 (7) | 2 (2)
Hemorrhage (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (General disorders) | 3 (3) | 8 (8)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Fever (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Blurred vision (Eye disorders) | 1 (1) | 4 (4)
Hyperglycemia (Endocrine disorders) | 1 (1) | 8 (8)
Gain weight (General disorders) | 0 (0) | 5 (5)
Infection (Infections and infestations) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days